CLINICAL TRIAL: NCT07339358
Title: Safety & Performance of the World Medica World Diverter Embolization Device
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: World Medica USA, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-001WM
Record Dates: First submitted 2026-01-12; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Intracranial Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- World Diverter Implantation (Experimental)
  Interventions: Device: Flow diverter implantation

INTERVENTIONS:
Device: Flow diverter implantation — Implantation of the World Diverter Embolization Device

SUMMARY:
The objective of this study is to investgiate the safety and clinical performance of the World Diverter Emoblization Device for the endovascular treatment of wide-neck (neck width ≥ 4 mm or dome-to-neck ratio <2) or fusiform intracranial aneurysms in the internal carotid artery (ICA) from the petrous segment to the terminus arising from a parent vessel with a diameter ≥ 2.5 mm and ≤ 5.5 mm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 22 to 80 years
* Subject, or subject's legal representative provided informed consent
* Subject agrees to the requirements of the study, including returning for required follow-up visits
* Parent artery diameter of 2.0-5.5 mm distal and proximal to the target IA
* Subject has a single target IA in the index procedure with the following characteristics: (1) Unruptured; (2) Located in the ICA from the petrous through the superior hypophyseal segments; and (3) Is a fusiform or saccular wide-necked IA with one of the following characteristics: (a) Small (< 5 mm) or medium (>5-10 mm) size with a neck width ≥ 4.0 mm or a dome-to-neck ratio of < 2; OR (b) Large (>10-25 mm) or giant (>25 mm) size

Exclusion Criteria:

* A subarachnoid or intracerebral hemorrhage in the 60 days preceding the index procedure
* A bleeding disorder or a platelet count of less than 100x103/mm3 or INR >1.5
* A contraindication to or inability to tolerate antiplatelet therapy
* An allergy to radiographic contrast agents
* An allergy to ￼ nickel, titanium, platinum, tungsten, or stainless steel
* An allergy to local or general anesthesia
* A history of untreated atrial fibrillation, untreated/uncontrollable hypertension, or other stroke risk factors
* A history of deep vein thrombosis or pulmonary embolism
* A history of heart failure, dilated cardiomyopathy, or congenital heart conditions
* Hypercoagulopathy or a hemorrhagic or coagulation deficiency refractory to medical therapy or subject refuses treatment with blood products
* Suffered a stroke within 180 days preceding the index procedure
* Had major surgery within the 30 days preceding or planned for the 180 days following the index procedure, including but not limited to intracranial stenting or coiling
* Target aneurysm has been previously treated with clipping, coiling, or flow diversion
* Had previous stenting of or implant in parent artery proximal to the target aneurysm that could interfere with delivery or performance of study device
* Asymptomatic extradural aneurysms requiring treatment
* Contraindication to computed tomography (CT) or magnetic resonance (MR)
* An unstable neurological deficit (i.e., worsening of a clinical condition within the 30 days preceding the index procedure)
* Evidence of an active systemic infection (including COVID-19) at index procedure
* Dementia or other cognitive condition limiting their ability to participate in the study
* A condition that may limit survival to less than 12 months post-index procedure
* Serum creatinine ≥2.5 mg/dL
* Had radiation or chemotherapy treatment either currently or within the 60 days preceding the index procedure
* Current enrollment in a separate clinical trial
* Another condition(s) that, in the opinion of the Investigator, could interfere with the ability to perform a safe or effective procedure
* Current pregnancy or plan to become pregnant within the 12 months following the index procedure, or be currently breastfeeding

Angiographic Exclusion Criteria:

* Anatomy not amenable to endovascular treatment, including but not limited to severe vessel tortuosity or stenosis
* Parent vessel stenosis is >50% in the target area
* Extracranial stenosis of the carotid artery >50%
* An intracranial mass
* More than one vessel segment requiring IA treatment in the 12 months following the index procedure
* Target aneurysm is mycotic or dissecting
* Target aneurysm is at bifurcation
* Target aneurysm will require coiling in addition to flow diversion, in Investigator's opinion

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety - Major Adverse Events (MAEs) | 12 months
  Composite incidence of the following events:
  * Major stroke (NIHSS increase of > 4) within 30 days post-procedure, defined as rapidly developing clinical signs of focal (or global) disturbance of cerebral function lasting > 24 hours with no apparent cause other than of vascular origin, including ischemic stroke or hemorrhagic stroke [i.e., intraparenchymal hemorrhage (IPH), subarachnoid hemorrhage (SAH), subdural hemorrhage (SDH), epidural hemorrhage (EDH)] accompanied with radiological evidence
  * Major ipsilateral stroke within 12 months post-procedure, defined as a major stroke (as defined above) occurring within the vascular distribution of the target artery
  * Neurological death within 12 months, defined as a death which directly resulted from a neurologic cause.
Primary Effectiveness - Complete Occlusion | 12 months
  The proportion of subjects with all of the following:
  * Complete (100%) occlusion of the target IA (Raymond-Roy Class I)
  * ≤ 50% stenosis of the parent artery at the target IA assessed by an independent Core Laboratory evaluation of angiography at 12 months post-procedure
  * No subsequent treatment of the target IA within 12 months post-procedure.

SECONDARY OUTCOMES:
Medium-Term Effectiveness | 6 months
  Complete IA occlusion
Medium-Term Parent Artery Stenosis | 6 months
  Parent Artery Stenosis
Medium-Term Functional Outcomes | 6 months
  Modified Rankin Score (0-6, 0=no symptoms, 6=dead) compared to baseline
Secondary Effectiveness - Adequate Occlusion | 12 months
  The proportion of subjects with all of the following:
  * Adequate occlusion of the target IA (Raymond-Roy Class I or II)
  * ≤ 50% stenosis of the parent artery at the target IA assessed by an independent Core Laboratory evaluation of angiography 12 months post-procedure
  * No subsequent treatment of the target IA within 12 months post-procedure
Long-Term Angiographic Outcome | 12 months
  Raymond-Roy IA classifications
Long-Term Parent Artery Stenosis | 12 months
  Parent Artery Stenosis
Long-Term Functional Outcome | 12 months
  Modified Rankin Score (0-6, 0=no symptoms, 6=dead) compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Tomasello, MD, Principal Investigator — Hospital Vall d'Hebron
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual participant data are protected by data privacy laws and are only provided for the purposes of this study following provision of participant informed consent.